CLINICAL TRIAL: NCT05019885
Title: A Pilot Study to Assess the Efficacy of Subanesthetic Doses of IV Ketamine in the Treatment Drug Resistant Epilepsy
Brief Title: The Efficacy of a Subanesthetic Doses of IV Ketamine in the Treatment Drug Resistant Epilepsy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Madeline Fields (Other)
Responsible Party: Sponsor-Investigator, Madeline Fields, Associate Professor of Neurology Co-Director Mount Sinai Epilepsy Center, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-20-01911
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Drug Resistant Epilepsy; Medically Refractory Epilepsy; Refractory Epilepsy
Keywords: drug resistant epilepsy; subanesthetic Ketamine hydrochloride
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Experimental clinical treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IV Ketamine Hydrochloride (Experimental): dose 0.5mg/kg of IV Ketamine Hydrochloride over 40 min
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Three times a week (M, W, F) for 2 consecutive weeks.

SUMMARY:
Ketamine is a medication that came into clinical practice in the 1960's. Ketamine is used as an anesthetic and to provide pain relief. Recently, Ketamine was approved to treat drug resistant depression using subanesthetic doses. In the hospital setting, intravenous anesthetic dosages are used to treat unrelenting seizures known as status epilepticus in comatose patients. Ketamine in subanesthetic doses has not been tried as a treatment for medication resistant seizures in the outpatient setting. This study would like to examine the effectiveness of subanesthetic ketamine in outpatients who suffer from drug resistant epilepsy.

DETAILED DESCRIPTION:
This is an open label pilot study that will evaluate the effectiveness of a sub-anaesthetic dose (0.5mg/kg) of IV Ketamine in Drug Resistant Epilepsy Patients. Mood assessments will also be administered. The study consists of 3 phases:

Screening : Seizure diary will be prospectively filled for 4 weeks and subjects must have at least 4 seizures in 28 days to proceed to the treatment phase. Baseline mood assessment will be performed (NDDI-E, QOLIE-10, GAD 7 )

Treatment Phase: This phase will consist of 6 study visits (3 visits/ week for 2 weeks). Patients will receive 0.5mg/kg Racemic ketamine IV over 40 min three times a week (M, W, F) for 2 consecutive weeks.

Treatment Visit 1: Monday Week 5(baseline seizures diary collected) Treatment Visit 2: Wednesday Week 5 Treatment Visit 3: Friday Week 5 Treatment Visit 4: Monday Week 6 Treatment Visit 5: Wednesday Week 6 Treatment Visit 6: Friday Week 6 (Mood assessments performed prior to infusion)

Post- Treatment Phase : This phase will consist of 5 post infusion safety assessments and 3 post-treatment assessments.

Post-Infusion Safety Assessment 1: Saturday Week 6 (Adverse Event Assessment) Post-Infusion Safety Assessment 2: Sunday Week 7 (Adverse Event Assessment) Post-Infusion Safety Assessment 3: Monday Week 7 (Adverse Event Assessment) Post-Infusion Safety Assessment 4: Monday Week 8 (Adverse Event Assessment) Post-Infusion Safety Assessment 5: Monday Week 9 (Adverse Event Assessment)

Post-Treatment Assessment 1: phone call week 10 (Seizure diary collection, mood assessments performed) Post-Treatment Assessment 2: phone call week 14 (Seizure diary) Post-Treatment Assessment 3: phone call week 18 (Seizure diary collection, mood assessments performed)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Adults (18 years or older)
* Cognitively impaired adults are not excluded (i.e. will be included in the study)
* Established diagnosis of Drug Resistant Epilepsy (DRE) i.e. failed two or more appropriately chosen anti-seizure medications (ASMs)
* EEG consistent with focal or generalized epilepsy
* Patients must have >4 focal aware, focal impaired aware, focal to bilateral tonic clonic or generalized tonic clonic seizures per month.
* Patients can be on >/= 1 anti-seizure medication (ASM) at the time of enrollment on stable doses 12 weeks prior to initiation
* Patients on Epilepsy devices: Vagal nerve stimulator (VNS), Deep brain stimulator (DBS) or Responsive Nerve Stimulator (RNS) must have remained stable for at least 4 weeks before the screening visit. Adjustment of devices is not allowed during the study.

Exclusion Criteria

* Patients <18 years of age
* Pregnant women
* Women that are breast feeding
* Patients who had >21 days of seizure freedom in the last year.
* Patients with a history of status epilepticus within 3 months of screening
* Patients with a history of alcoholism of drug misuse within the last 2 years
* Unstable medical illness
* Serious or imminent suicidal or homicidal risk
* Patients with cardiovascular disease
* Patients with schizophrenia
* Patients with history of aneurysm or aortic dissection, arteriovenous malformation and intracerebral hemorrhage
* Patients that are immobile i.e. wheel chair bound, bed ridden individuals
* Patients on psychostimulants (amphetamines, methylphenidate etc.) and Monoamine oxidase inhibitors (selegiline, isocarboxazid, phenelzine etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with seizure reduction | 2 week during active treatment
  50% seizure reduction during the 2 week period of active treatment
Number of participants with seizure reduction | 28 days post infusion
  50% seizure reduction during the 28 days post-infusion.
Seizure frequency | 3 months post infusion
  Return to pre-ketamine infusion seizure frequency in 3 months

SECONDARY OUTCOMES:
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) Score | Week 6
  The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) is a 6-item questionnaire validated to screen for depression in people with epilepsy. Scores range from 6 - 24, with higher scores indicating more depressive symptoms.
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) Score | Week 10
  The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) is a 6-item questionnaire validated to screen for depression in people with epilepsy. Scores range from 6 - 24, with higher scores indicating more depressive symptoms.
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) Score | Week 14
  The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) is a 6-item questionnaire validated to screen for depression in people with epilepsy. Scores range from 6 - 24, with higher scores indicating more depressive symptoms.
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) Score | Week 18
  The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) is a 6-item questionnaire validated to screen for depression in people with epilepsy. Scores range from 6 - 24, with higher scores indicating more depressive symptoms.
Quality of Life in Epilepsy (QOLIE-10) | Week 6
  Quality of Life in Epilepsy (QOLIE)-10 scale is a validated, reliable instrument measuring quality of life on a scale from 10-51, lower score indicates better health outcome.
Quality of Life in Epilepsy (QOLIE-10) | Week 10
  Quality of Life in Epilepsy (QOLIE)-10 scale is a validated, reliable instrument measuring quality of life on a scale from 10-51, lower score indicates better health outcome.
Quality of Life in Epilepsy (QOLIE-10) | Week 14
  Quality of Life in Epilepsy (QOLIE)-10 scale is a validated, reliable instrument measuring quality of life on a scale from 10-51, lower score indicates better health outcome.
Quality of Life in Epilepsy (QOLIE-10) | Week 18
  Quality of Life in Epilepsy (QOLIE)-10 scale is a validated, reliable instrument measuring quality of life on a scale from 10-51, lower score indicates better health outcome.
General Anxiety Disorder 7-item questionnaire (GAD-7) | week 6
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms.
General Anxiety Disorder 7-item questionnaire (GAD-7) | week 10
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms.
General Anxiety Disorder 7-item questionnaire (GAD-7) | week 14
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms.
General Anxiety Disorder 7-item questionnaire (GAD-7) | week 18
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Madeline Fields, MD, Principal Investigator — Icahn School of Medicine; Lara Marcuse, MD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Undecided at this time

REFERENCES:
- [Background] aan het Rot M, Collins KA, Murrough JW, Perez AM, Reich DL, Charney DS, Mathew SJ. Safety and efficacy of repeated-dose intravenous ketamine for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):139-45. doi: 10.1016/j.biopsych.2009.08.038. PMID 19897179
- [Background] Aram JA, Martin D, Tomczyk M, Zeman S, Millar J, Pohler G, Lodge D. Neocortical epileptogenesis in vitro: studies with N-methyl-D-aspartate, phencyclidine, sigma and dextromethorphan receptor ligands. J Pharmacol Exp Ther. 1989 Jan;248(1):320-8. PMID 2536430
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Brodie MJ. Road to refractory epilepsy: the Glasgow story. Epilepsia. 2013 May;54 Suppl 2:5-8. doi: 10.1111/epi.12175. PMID 23646962
- [Background] Dingledine R, Borges K, Bowie D, Traynelis SF. The glutamate receptor ion channels. Pharmacol Rev. 1999 Mar;51(1):7-61. No abstract available. PMID 10049997
- [Background] Esaian D, Joset D, Lazarovits C, Dugan PC, Fridman D. Ketamine continuous infusion for refractory status epilepticus in a patient with anticonvulsant hypersensitivity syndrome. Ann Pharmacother. 2013 Nov;47(11):1569-76. doi: 10.1177/1060028013505427. Epub 2013 Oct 9. PMID 24259603
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Fujikawa DG. Neuroprotective effect of ketamine administered after status epilepticus onset. Epilepsia. 1995 Feb;36(2):186-95. doi: 10.1111/j.1528-1157.1995.tb00979.x. PMID 7821277
- [Background] Hsieh CY, Sung PS, Tsai JJ, Huang CW. Terminating prolonged refractory status epilepticus using ketamine. Clin Neuropharmacol. 2010 May;33(3):165-7. doi: 10.1097/WNF.0b013e3181d1e3cd. PMID 20098301
- [Background] Kramer AH. Early ketamine to treat refractory status epilepticus. Neurocrit Care. 2012 Apr;16(2):299-305. doi: 10.1007/s12028-011-9668-7. PMID 22237581
- [Background] Kramer U, Shorer Z, Ben-Zeev B, Lerman-Sagie T, Goldberg-Stern H, Lahat E. Severe refractory status epilepticus owing to presumed encephalitis. J Child Neurol. 2005 Mar;20(3):184-7. doi: 10.1177/08830738050200030301. PMID 15832606
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Gaspard N, Foreman B, Judd LM, Brenton JN, Nathan BR, McCoy BM, Al-Otaibi A, Kilbride R, Fernandez IS, Mendoza L, Samuel S, Zakaria A, Kalamangalam GP, Legros B, Szaflarski JP, Loddenkemper T, Hahn CD, Goodkin HP, Claassen J, Hirsch LJ, Laroche SM. Intravenous ketamine for the treatment of refractory status epilepticus: a retrospective multicenter study. Epilepsia. 2013 Aug;54(8):1498-503. doi: 10.1111/epi.12247. Epub 2013 Jun 12. PMID 23758557
- [Background] Lang E, Mallien AS, Vasilescu AN, Hefter D, Luoni A, Riva MA, Borgwardt S, Sprengel R, Lang UE, Gass P, Inta D. Molecular and cellular dissection of NMDA receptor subtypes as antidepressant targets. Neurosci Biobehav Rev. 2018 Jan;84:352-358. doi: 10.1016/j.neubiorev.2017.08.012. Epub 2017 Aug 23. PMID 28843752
- [Background] Lapidus KA, Levitch CF, Perez AM, Brallier JW, Parides MK, Soleimani L, Feder A, Iosifescu DV, Charney DS, Murrough JW. A randomized controlled trial of intranasal ketamine in major depressive disorder. Biol Psychiatry. 2014 Dec 15;76(12):970-6. doi: 10.1016/j.biopsych.2014.03.026. Epub 2014 Apr 3. PMID 24821196
- [Background] Lawn ND, Bamlet WR, Radhakrishnan K, O'Brien PC, So EL. Injuries due to seizures in persons with epilepsy: a population-based study. Neurology. 2004 Nov 9;63(9):1565-70. doi: 10.1212/01.wnl.0000142991.14507.b5. PMID 15534237
- [Background] McCagh J, Fisk JE, Baker GA. Epilepsy, psychosocial and cognitive functioning. Epilepsy Res. 2009 Sep;86(1):1-14. doi: 10.1016/j.eplepsyres.2009.04.007. Epub 2009 Jul 18. PMID 19616921
- [Background] Lent JK, Arredondo A, Pugh MA, Austin PN. Ketamine and Treatment-Resistant Depression. AANA J. 2019 Oct;87(5):411-419. PMID 31612847
- [Background] Mazarati AM, Wasterlain CG. N-methyl-D-asparate receptor antagonists abolish the maintenance phase of self-sustaining status epilepticus in rat. Neurosci Lett. 1999 Apr 23;265(3):187-90. doi: 10.1016/s0304-3940(99)00238-4. PMID 10327162
- [Background] Mewasingh LD, Sekhara T, Aeby A, Christiaens FJ, Dan B. Oral ketamine in paediatric non-convulsive status epilepticus. Seizure. 2003 Oct;12(7):483-9. doi: 10.1016/s1059-1311(03)00028-1. PMID 12967577
- [Background] Mohanraj R, Norrie J, Stephen LJ, Kelly K, Hitiris N, Brodie MJ. Mortality in adults with newly diagnosed and chronic epilepsy: a retrospective comparative study. Lancet Neurol. 2006 Jun;5(6):481-7. doi: 10.1016/S1474-4422(06)70448-3. PMID 16713919
- [Background] Murrough JW, Burdick KE, Levitch CF, Perez AM, Brallier JW, Chang LC, Foulkes A, Charney DS, Mathew SJ, Iosifescu DV. Neurocognitive effects of ketamine and association with antidepressant response in individuals with treatment-resistant depression: a randomized controlled trial. Neuropsychopharmacology. 2015 Mar 13;40(5):1084-90. doi: 10.1038/npp.2014.298. PMID 25374095
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761
- [Background] Niciu MJ, Ionescu DF, Richards EM, Zarate CA Jr. Glutamate and its receptors in the pathophysiology and treatment of major depressive disorder. J Neural Transm (Vienna). 2014 Aug;121(8):907-24. doi: 10.1007/s00702-013-1130-x. Epub 2013 Dec 8. PMID 24318540
- [Background] Pruss H, Holtkamp M. Ketamine successfully terminates malignant status epilepticus. Epilepsy Res. 2008 Dec;82(2-3):219-22. doi: 10.1016/j.eplepsyres.2008.08.005. Epub 2008 Sep 19. PMID 18804344
- [Background] Rosati A, De Masi S, Guerrini R. Ketamine for Refractory Status Epilepticus: A Systematic Review. CNS Drugs. 2018 Nov;32(11):997-1009. doi: 10.1007/s40263-018-0569-6. PMID 30232735
- [Background] Tarocco A, Ballardini E, Garani G. Use of ketamine in a newborn with refractory status epilepticus: a case report. Pediatr Neurol. 2014 Jul;51(1):154-6. doi: 10.1016/j.pediatrneurol.2014.03.006. Epub 2014 Mar 15. PMID 24938144
- [Background] Scott AJ, Sharpe L, Hunt C, Gandy M. Anxiety and depressive disorders in people with epilepsy: A meta-analysis. Epilepsia. 2017 Jun;58(6):973-982. doi: 10.1111/epi.13769. Epub 2017 May 3. PMID 28470748
- [Background] Sheth RD, Gidal BE. Refractory status epilepticus: response to ketamine. Neurology. 1998 Dec;51(6):1765-6. doi: 10.1212/wnl.51.6.1765. No abstract available. PMID 9855547
- [Background] Synowiec AS, Singh DS, Yenugadhati V, Valeriano JP, Schramke CJ, Kelly KM. Ketamine use in the treatment of refractory status epilepticus. Epilepsy Res. 2013 Jul;105(1-2):183-8. doi: 10.1016/j.eplepsyres.2013.01.007. Epub 2013 Jan 29. PMID 23369676
- [Background] Ubogu EE, Sagar SM, Lerner AJ, Maddux BN, Suarez JI, Werz MA. Ketamine for refractory status epilepticus: a case of possible ketamine-induced neurotoxicity. Epilepsy Behav. 2003 Feb;4(1):70-5. doi: 10.1016/s1525-5050(02)00643-1. PMID 12609230
- [Background] Walker MC, Howard RS, Smith SJ, Miller DH, Shorvon SD, Hirsch NP. Diagnosis and treatment of status epilepticus on a neurological intensive care unit. QJM. 1996 Dec;89(12):913-20. doi: 10.1093/qjmed/89.12.913. PMID 9015485
- [Background] Yeh PS, Shen HN, Chen TY. Oral ketamine controlled refractory nonconvulsive status epilepticus in an elderly patient. Seizure. 2011 Nov;20(9):723-6. doi: 10.1016/j.seizure.2011.06.001. Epub 2011 Jul 2. PMID 21724423
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Zeiler FA, Kaufmann AM, Gillman LM, West M, Silvaggio J. Ketamine for medically refractory status epilepticus after elective aneurysm clipping. Neurocrit Care. 2013 Aug;19(1):119-24. doi: 10.1007/s12028-013-9858-6. PMID 23702695
- [Background] Zeiler FA, Teitelbaum J, Gillman LM, West M. NMDA antagonists for refractory seizures. Neurocrit Care. 2014 Jun;20(3):502-13. doi: 10.1007/s12028-013-9939-6. PMID 24519081